CLINICAL TRIAL: NCT02664051
Title: The Role of Mast Cells on Duodenal Permeability After Duodenal Acid Perfusion in Healthy Volunteers
Brief Title: Mast Cells in Acid-induced Intestinal Permeability
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inactive
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: S56881; 2015-000244-42 (EudraCT Number)
Record Dates: First submitted 2015-11-24; First posted 2016-01-26 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2015-11

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — Cromolyn Sodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): mannitol
  Interventions: Drug: placebo
- disodium cromoglycate (Active Comparator): disodium cromoglycate
  Interventions: Drug: Nalcrom

INTERVENTIONS:
Drug: Nalcrom — Drug: disodium cromoglycate 100mg 4x2 daily
  Other Names:
  • Nalcrom
  Arms: disodium cromoglycate
Drug: placebo — 100mg 4x2 daily mannitol
  Arms: placebo

SUMMARY:
This is a randomized, double-blind, cross-over study in healthy volunteers. In the first part, the duodenum of the participants will be perfused with acid or saline, during which intragastric pressure will be monitored to assess activation of the duodenogastric reflex. After perfusion, duodenal biopsies will be collected to evaluate mucosal integrity. In the second part, healthy volunteers are treated with the mast cell stabilizer disodium cromoglycate or with a placebo during 14 days. Subsequently, the duodenum will be perfused with acid and intragastric pressure and mucosal integrity will be evaluated.

DETAILED DESCRIPTION:
Despite intensive research, the pathophysiology of functional dyspepsia remains unknown. The investigators recently demonstrated that functional dyspepsia patients display impaired duodenal mucosal integrity and low-grade mucosal inflammation. As studies have also shown that functional dyspepsia patients present with an increased spontaneous duodenal acid exposure, the hypothesis of this study is that increased duodenal acid exposure results in increased duodenal permeability via mast cell activation. This will also induce activation of the duodenogastric reflex, resulting in gastric relaxation, eventually leading to the generation of dyspeptic symptoms. The general aim of this project is to assess the effect of mast cell inhibition on duodenal mucosal integrity and intragastric pressure of healthy volunteers after acid infusion in the duodenum.

The study will be a randomized, double-blind, cross-over study in 20 healthy volunteers and consists of 2 parts. (1) In the first part, 10 healthy volunteers will be perfused with acid (0.1N HCl) or 0.9% saline during 30 minutes at a rate of 5 mL/min with an interval of at least one month. During acid/saline perfusion, intragastric pressure will be measured with a high resolution manometry system to evaluate activation of the duodenogastric reflex. Dyspeptic symptoms will be scored 1 minute before and every 5 minutes during the infusion. After perfusion, endoscopy will be performed and duodenal biopsies will be obtained to evaluate mucosal integrity using Ussing chambers and by assessing the expression of cell-to-cell adhesion proteins (real-time PCR, immunofluorescence and western blot). (2) In the second part, 10 healthy volunteers will be perfused with acid after a placebo treatment and after treatment with the mast cell stabilizer disodium cromoglycate 100mg 4x2/day (with an interval of at least one month). The rest of the study continues as described in part 1.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* - refused informed consent
* pregnant women or women who are breastfeeding
* symptoms or history of gastrointestinal disease
* diabetes mellitus
* coagulation disorders/anticoagulant therapy
* first degree relatives with celiac disease, Crohn's disease or type I diabetes mellitus
* taking antihistamines, ketotifen, cromoglycate, acetylsalicylates, NSAIDs, anticholinergics, theophylline, β2-agonists, codeine or opioid derivatives 2 weeks prior to the study
* taking steroid or immunosuppressive drugs 6 months prior to the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
evaluation of transepithelial resistance (mucosal integrity) of duodenal biopsies after duodenal saline or acid perfusion, after treatment with placebo or a mast cell stabilizer | 2 weeks

SECONDARY OUTCOMES:
evaluation of intragastric pressure during duodenal saline or acid perfusion, after treatment with placebo or a mast cell stabilizer | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Translational Research Center for Gastrointestinal Disorders (TARGID), KU Leuven Campus Gasthuisberg O&N1, Leuven, Vlaams Brabant, Belgium